CLINICAL TRIAL: NCT02632318
Title: Dawn Simulation as a Passive Countermeasure to Postural Hypotension in Healthy Older Adults
Brief Title: Dawn Simulation and Postural Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Velux Fonden (Other); Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Assistant Professor, VA Palo Alto Health Care System
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-36269
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Light (Experimental): Dawn simulation for 30 minutes prior to habitual wake time
  Interventions: Device: Light
- No light (No Intervention): Darkness for 30 minutes prior to habitual wake time

INTERVENTIONS:
Device: Light — 30 minutes of dawn simulation
  Arms: Light

SUMMARY:
One of the most physiologically demanding things that older people do every day is to get up in the morning. After spending a night laying flat, where the blood distributes evenly across the body, when they stand in the morning (and the blood rushes to their feet), their cardiovascular system may not be able to compensate and maintain blood flow to the brain. This phenomenon is known as orthostatic or postural hypotension. The investigators have found in a group of young individuals that use of a dawn-simulation light that gradually wakes the brain is able to increase cardiovascular tone prior to arising. The goal of this experiment is to determine whether this dawn simulation light is able to increase cardiovascular tone in older adults such that they would have reduced or absent postural hypotension when they awaken in the morning. This would greatly reduce the risks of falls and their associated morbidities in older adults.

ELIGIBILITY:
Inclusion Criteria:

* History of falls or dizziness at exit from bed in the morning (at least two incidents in the past year)
* At least 20/200 corrected visual acuity
* Stable health
* Normal hearing

Exclusion Criteria:

* Regular cigarette smoker
* Alcohol abuse
* Drug abuse

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Sympathovagal balance derived from blood pressure measurement | 30 minutes
  measure of sympathovagal balance derived from blood pressure measurement at wake time

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data will be made available upon request following publication of summary data.

REFERENCES:
- [Derived] Gabel V, Miglis M, Zeitzer JM. Effect of artificial dawn light on cardiovascular function, alertness, and balance in middle-aged and older adults. Sleep. 2020 Oct 13;43(10):zsaa082. doi: 10.1093/sleep/zsaa082. PMID 32307533